CLINICAL TRIAL: NCT03021031
Title: Circuit-Based Deep Brain Stimulation for Parkinson's Disease; Udall Clinical Core
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEURO-2016-25066
Record Dates: First submitted 2017-01-09; First posted 2017-01-13 (Estimated); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

INTERVENTIONS:
Other: Observational — Observational study

SUMMARY:
The goal of this project is to provide comprehensive longitudinal assessments of a cohort of PD patients before, during, and after DBS surgery, including neurological, neurophysiological, and neuropsychological data.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* Diagnosis of Parkinson's disease
* Candidate for DBS

Exclusion Criteria:

* Diagnosis of dementia
* Pregnant women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with Parkinson's Disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Registry | 5 Years
  This is a registry of patients undergoing DBS surgery. The goal of this project is to provide comprehensive longitudinal assessments of a cohort of PD patients before, during, and after DBS surgery, including neurological, neurophysiological, and neuropsychological data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States